CLINICAL TRIAL: NCT04899687
Title: Fluoxetine/Dextromethorphan in Obsessive-Compulsive and Related Disorders: an Open-Label Crossover Pilot Study
Brief Title: Study of Dextromethorphan in OCD and Related Disorders
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Avy L. & Roberta L. Miller Foundation (Unknown)
Responsible Party: Principal Investigator, Peter J van Roessel, MD PhD, Clinical Associate Professor, Stanford University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 60569
Record Dates: First submitted 2021-05-13; First posted 2021-05-24 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Obsessive-Compulsive Disorder; Illness Anxiety Disorder; Body Dysmorphic Disorders; Somatic Symptom Disorder
Keywords: OCD; BDD; IAD; SSD; Fluoxetine; Dextromethorphan
MeSH Terms: conditions — Obsessive-Compulsive Disorder; Body Dysmorphic Disorders | interventions — Fluoxetine; Dextromethorphan

STUDY DESIGN:
Intervention Model Description: After signing consent and baseline assessments, participants will be randomized 1:1 to Group A or Group B for the purposes of sequencing fluoxetine vs combined fluoxetine/dextromethorphan treatment periods.
Who Masked: Outcomes Assessor
Masking Description: Symptom rating will be done by independent evaluators blind to treatment allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Group A: fluoxetine then fluoxetine plus dextromethorphan (Experimental): Group A participants will take fluoxetine 20mg (or prior dose) daily for 4 weeks, and will then continue fluoxetine while adding over the counter dextromethorphan, with doses increasing weekly as tolerated, for 4 weeks.
  Interventions: Drug: Fluoxetine; Drug: Dextromethorphan
- Group B: fluoxetine plus dextromethorphan then fluoxetine (Experimental): Group B participants will take fluoxetine 20mg (or prior dose) daily together with over the counter dextromethorphan, with doses increasing weekly as tolerated, for 4 weeks, and then will stop dextromethorphan, continuing fluoxetine alone for 4 weeks.
  Interventions: Drug: Fluoxetine; Drug: Dextromethorphan

INTERVENTIONS:
Drug: Fluoxetine — Fluoxetine 20mg (or previously prescribed dose) will be taken once daily by mouth for 8 weeks
  Other Names: Prozac
Drug: Dextromethorphan — Dextromethorphan, an over-the-counter cough suppressant, will be taken by mouth twice daily for four weeks of the study, starting at 15mg per dose, and increasing weekly as tolerated to a maximum of 60mg per dose.

SUMMARY:
The purpose of the study is to assess the tolerability and efficacy of dextromethorphan in combination with fluoxetine for symptom relief in OCD and related disorders.

DETAILED DESCRIPTION:
Obsessive compulsive disorder (OCD) and the related disorders body dysmorphic disorder (BDD), somatic symptom disorder (SSD) and illness anxiety disorder (IAD) are psychiatric conditions characterized by recurrent, intrusive thoughts, feelings or images (obsessions or preoccupations) and repetitive or ritualized behaviors or avoidance performed to relieve obsession or preoccupation-related anxiety. They are a significant cause of mental health-related disability, and are inadequately served by available treatments.

This study tests whether an over-the-counter cough suppressant medicine, dextromethorphan, may offer symptom relief when combined with a low dose of fluoxetine, a standard prescription treatment for OCD and related disorders.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of obsessive-compulsive disorder (OCD), body dysmorphic disorder (BDD), illness anxiety disorder (IAD) or somatic symptom disorder (SSD)
* Living within California
* Capacity to provide informed consent

Exclusion Criteria:

* Current bipolar disorder or psychotic disorder
* Active moderate or severe substance use disorder, lifetime severe substance use disorder
* Pregnant or nursing women
* Use of prescribed psychotropic medications other than fluoxetine for 2 weeks prior to study start
* Having commenced OCD-targeted exposure and response-prevention (ExRP) psychotherapy within 2 months of study start

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-01-20 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Improvement in OCD or related disorder symptoms as measured by the Y-BOCS | Change from baseline will be assessed at 4 weeks and at 8 weeks.
  Improvement in OCD severity is measured by the Yale-Brown Obsessive Compulsive Scale (Y-BOCS), a gold standard measure of the severity of obsessions and compulsions. Variants of the Y-BOCS designed for assessment of body dysmorphic disorder or illness anxiety disorder/somatic symptom disorder will be used as appropriate. Y-BOCS scores range from 0 to 40, with higher scores indicating greater severity of symptoms. Response will be defined as a 35% reduction in Y-BOCS score.

SECONDARY OUTCOMES:
Improvement in clinical insight as measured by the BABS | Change from baseline will be assessed at 4 weeks and at 8 weeks.
  Improvement in clinical insight is measured by the Brown Assessment of Beliefs Scale (BABS), a scale assessing multiple dimensions of clinical insight as relevant to OCD and related disorders. The BABS rates multiple dimensions of clinical insight related to an identified belief. BABS scores range from 0-24, with higher scores indicating greater insight impairment. Response will be defined as a 35% reduction in BABS score.

CONTACTS AND LOCATIONS:
Overall Officials: Peter J van Roessel, MD PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No